CLINICAL TRIAL: NCT04434235
Title: Effects of Additional Axial Load on Cervical Motor Control
Acronym: Axial
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00830
Record Dates: First submitted 2020-04-28; First posted 2020-06-16 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: cervical spine
MeSH Terms: interventions — Weight-Bearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dynamic cervical stability: The participant is asked to move the head in 6 directions in a sitting position and 30° leaning backward sitting position; lateral flexion (left / right), flexion, extension, and rotation (left / right). Results are to be taken for each direction and random at each axial load-level (0 kg, 1kg, 2 kg, and 3 kg). In total 24 measurements.
  The duration of all measurement will be 60 minutes.
  Interventions: Other: axial load
- Cervical Stiffness: The participant is asked to move the head in 4 directions; flexion, extension, and rotation (left / right). Joint-Position Error measurements will be executed in neutral sitting position. Additionally, stiffness will be measured in neutral sitting position and neutral sitting position with 45° cervical flexion. All measurements will be performed with 0 kg and 3 kg axal loading. In total 18 measurements.The duration of all measurement will be 60 minutes.
  Interventions: Other: axial load

INTERVENTIONS:
Other: axial load — With a helmet with Velcro fastener we will add additional weight to produce axial load on the cervical spine

SUMMARY:
he objective of this study is to examine the influence of additional axial load abd body position on cervical motor control in young healthy adults.

DETAILED DESCRIPTION:
Motor control of the cervical spine is impotent for responsible for maintaining balance during daily living activities and to withstand external loads. Stabilization-aspects of the cervical spine is very complex, passive (ligaments, joint capsule and the skin and active (muscles), and neurological subsystems are involved. Mostly proprioceptive testing and exercises like head and neck position sense testing and re-training have been an integral part of rehabilitation. Another method to evaluate spinal motor control is the assessment of spinal stiffness. The main objective of this study is to explore the effects of additional axial loading on motion control in healthy individuals. Does the motor control of the cervical spine in healthy subjects change with additional axial load or body position? A better understanding of spinal stiffness and neck position sense leads to novel insights into spinal cervical stabilization mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Healthy participant's Signed informed consent after being informed

Exclusion Criteria:

Acute pain Chronic neck pain Undergone Neck surgery Neck Disability Index Score > 15

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change of neck joint-position error between differnent weight conditions | 20 minutes group cervical stiffness
  Joint-position error will be will be assessed with Sensomove. It consists of the 3D senscoordination sensor, an adjustable headband, and basic software for motion feedback of head movements. The change of Joint-Position Error with and without additional axial load will be assessed.
Change of neck joint-position error between two sitting positions | 20 minutes group Dynamic cervical stability
  Joint-position error will be will be assessed with Sensomove It consists of the 3D senscoordination sensor, an adjustable headband, and basic software for motion feedback of head movements. The change of Joint-Position Error with axial load (3kg) between two sitting positions will be assessed.
Change of neck range of motion between different weight conditions | 20 minutes group cervical stiffness
  Range of motion will be will be assessed with Sensomove It consists of the 3D senscoordination sensor, an adjustable headband, and basic software for motion feedback of head movements. The change of Rage of motion with and without additional axial load will be assessed.
Change of spinal stiffness between different sitting positions and loading conditions | 20 minutes group cervical stiffness
  The device measures tissue compliance according to the concept of impulse-response. A force of exact 20 Newton will be applied from the device to the process spinous. The expected impulse-response (result) will be between 20 Newton and 40 Newton. The change of spinal stiffness due sitting position and loading will be assessed.

SECONDARY OUTCOMES:
Pain during measuring | 2 minutes
  The visual analogue scale will be used to quantify pain, if any of the measurements is painful. The participant is asked to rate his pain intensity on a straight line (100mm) with two endpoints.
Self-administered neck mobility | 4 minutes
  Self-administered neck mobility questionnaire is a self-administered questionnaire that uses visual analog scales to measure pain-free active rage of motion for all neck movements. The patient is asked to place a mark on a 100 mm line (0 mm = "no movement possible" and 100 mm = "as far as possible"). The total score is the sum of the individual scores (min. score (600) = no restrictions and max. score (0) = total restriction)
Neck Disability Index | 4 minutes
  The Neck Disability Index is a self-report questionnaire with 10-items: pain intensity, personal care, lifting, work, headaches, concentration, sleeping, driving, reading, and recreation. The response to each item is rated on a 6-point scale from 0 (no disability) to 5 (complete disability). The numeric responses for each item are summed for a total score ranging between 0 and 50.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No